CLINICAL TRIAL: NCT06809205
Title: Efficacy and Safety of Tadalafil, Tamsulosin, and Their Combinations in Treating Lower Urinary Tract Symptoms in BPH Patients with Prostate Volumes ≤ 40 Ml: a Prospective Comparative Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Dogha, lecturer of urology- faculty of medicine- fayoum university, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R 450
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: BPH with Other Lower Urinary Tract Symptoms
Keywords: Tamsulosin, tadalafil, BPH and LUTS
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Group A was administered Tamsulosin (0.4 mg per day)
  Interventions: Drug: Tamsulosin 0.4 mg
- Group B (Experimental): Group B was administered tadalafil (5 mg per day)
  Interventions: Drug: Tadalafil 5mg
- group c (Experimental): administered tadalafil and tamsulosin 0.4 mg
  Interventions: Drug: Tamsulosin and Tadalafil

INTERVENTIONS:
Drug: Tamsulosin 0.4 mg — administered tamsulosin 0.4 mg
  Other Names: group A
  Arms: Group A
Drug: Tadalafil 5mg — administered tadalafil 5 mg
  Other Names: group B
  Arms: Group B
Drug: Tamsulosin and Tadalafil — administered tamsulosin 0.4 mg plus tadalafil 5 mg
  Other Names: Group C
  Arms: group c

SUMMARY:
Abstract:

Objective: To examine the influence of tadalafil and tamsulosin versus their combinations in the treatment of lower urinary tract symptoms in mildly enlarged prostates below 40 ml in volume.

Materials and methods: A prospective randomized study was done at Fayoum and Beni-Suef University Hospitals in Egypt from December 2022 to August 2023. A total of 95 male participants aged over 45 years, all presenting with mild to intense lower urinary tract symptoms, were enrolled. Participants were randomized into three groups: Group A was administered Tamsulosin (0.4 mg per day), Group B was administered tadalafil (5 mg per day), and Group C was administered a mixture of both medications. The study assessed multiple parameters, the primary endpoint parameter was the International Prostate Symptom Score (IPSS) and the other secondary parameters were the five-item International Index of Erectile Function (IIEF-5), maximum urinary flow rate (Q-max), post-void residual urine (PVR), and the quality of life (QoL). At baseline, these parameters were assessed, followed by evaluations at 1, 3, and 6 months after treatment.

Key words. Tamsulosin, tadalafil, BPH and LUTS.

DETAILED DESCRIPTION:
Efficacy and Safety of Tadalafil, Tamsulosin, and Their Combinations in Treating Lower Urinary Tract Symptoms in BPH Patients with Prostate Volumes ≤ 40 ml: A Prospective Comparative Study.

Mohamed Mahmoud Dogha*1, Mahmoud Shoukry ElAdawy¹, Rabie M Ibrahim², Ahmed Yousef2, ,Samia Heikal3, Mahmoud AbdElhamid4, Ahmed Abdalgalil1, Hossam Shaker¹.

1. Department of Urology, Faculty of Medicine, Fayoum University, Egypt
2. Department of Urology, Faculty of Medicine, Beni-suef University, Egypt
3. Diagnostic Radiology Department, National Cancer Institute, Cairo University
4. Department of Urology, Faculty of Medicine, Cairo University, Egypt

   *Email: mma16@fayoum.edu.eg

   Introduction:

   Lower urinary tract symptoms (LUTS) are frequently triggered by benign prostatic enlargement (BPE), such as storage symptoms like nocturia, frequency, and urgency, along with voiding symptoms like hesitancy, weak flow, and straining, all of which can substantially impact the total quality of life for a patient. [1, 2] Treatment options for LUTS related to BPE include surgical intervention, pharmacotherapy (such as 5-alpha reductase inhibitors, phosphodiesterase 5 inhibitors, alpha blockers, and phytotherapies) and other approaches. [3, 4] alpha blockers work by reducing prostate tone through the inhibition of noradrenaline's influence on smooth muscle cells in the prostate. [5] Although the complete clinical effects of alpha blockers may take a few weeks to become evident, notable improvements can often be seen within hours to days. [6] These medications are effective in alleviating both storage and voiding LUTS without reducing prostate size, although they tend to be more effective in patients with a prostate size of lower than 40 ml. [7-10] Despite these advancements in the Qmax and the IPSS can be sustained for at least four years with alpha blocker therapy. phosphodiesterase 5 inhibitors reduce smooth muscle tone in the urethra, prostate, and detrusor, and their chronic use may raise oxygenation, and blood flow, and potentially diminish chronic inflammation in the lower urinary tract. However, the precise way in which they influence LUTS is still not well understood. [11-13] Our study aimed to examine the efficacy of tamsulosin versus tadalafil, and their combination; in treating LUTS/BPE in individuals with a prostate size ≤ 40 ml.

   Materials and methods:

   Our prospective randomized clinical assessment was performed from December 2022 to August 2023 at the Urology Department of Fayoum and Beni-suef University Hospitals Randomization was carried out using a sealed envelope method. The Review Board, an ethical commission, received approval (approval number: R 450) from the hospital ethics committee at the Fayoum University Faculty of Medicine. After receiving a detailed explanation of the study's objectives, participants were made aware of the purpose and benefits of the analysis. The participants in the study provided their consent willingly. Moreover, written consent was secured in advance. The confidentiality of the information collected was assured to the participants. Inclusion criteria were male patients aged ≥ 45years with prostate volume less than 40 ml, with mild to intense LUTS/BPH as regard to IPSS.The exclusion criteria included a prostate-specific antigen (PSA) level exceeding 4 ng/mL, a prostate volume exceeding 40 ml, an amount of remaining urine of 300 mL or more, the utilize of 5-alpha reductase inhibitors (5-ARIs) in the past three months, a history of prostate surgery or malignancy, urethral stricture, urinary retention, bladder stones, neurological diseases affecting bladder function, cardiovascular diseases, and treatment with nitrates. Patients were divided into three groups: group A was administered 0.4 mg tamsulosin per day, group B was administered tadalafil 5mg daily, and group C was administered a mixture of both tadalafil and tamsulosin. Each patient underwent assessments at four distinct intervals: at presentation and after 1, 3, and 6 months of treatment. At the initial presentation, comprehensive assessments were performed, while follow-up visits included evaluations of the IIEF-5, IPSS, uroflowmetry, PVR and IPSS QoL scores. The results from the three groups were recorded at all four visits and subsequently compared and analyzed statistically.All ultrasounds were performed by the same radiologist to eliminate the bias of different radiology operators Statistical methods: G * power was used to determine a minimum sample size of 90. The target sample size was computed with an alpha value of 0.05, an effect size of 0.25, and a power of study of 0.8. The data were analyzed using SPSS (Statistical Package for the Social Sciences) version 28 (IBM Corp., Armonk, NY, USA). The mean and standard deviation of the data served as a summary. Groups were compared using analysis of variance (ANOVA), followed by a post-hoc multiple comparisons test (Chan, 2003). Data was double checked for normality using normality plots and Shapiro Wilk test and proved not to be deviated from normal distribution. According to [14], statistical significance was defined as a p-value less than 0.05.

   Declarations Ethics approval and consent to participate: The Review Board, an ethical commission, received approval (approval number: R 450) from the hospital ethics committee at the Fayoum University Faculty of Medicine in accordance with the declaration of Helsinki. And every participant provided a cleared and detailed consent.

   Conflict of Interest: None. Funding: None.

   Authors' contributions:

   Mohamed Mahmoud Dogha conducted conception and design of the study. Mahmoud S. ElAdawy and Mahmoud AbdElhamid performed interpretation of data, work design. Hossam shaker, Samia Heikal and Ahmed Abdalgalil did conception and design of the study, drafted the manuscript, interpretation of data. Rabie M. Ibrahim and Ahmed Yousif drafted the manuscript, Data analysis

   Abbreviations:
5. ARIs: 5-alpha reductase inhibitors BPE: Benign prostatic enlargement IEFF-5: International Index of Erectile Function 5 items IPSS: international prostate symptom score LUTS: Lower urinary tract symptoms PDE5Is: phosphodiesterase type 5 inhibitors PSA: Prostate-specific antigen Qmax: maximum urinary flow rate QoL: quality of life

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were male patients aged ≥ 45years with prostate volume less than 40 ml, with mild to intense LUTS/BPH as regard to IPSS.

Exclusion Criteria:

* The exclusion criteria included a prostate-specific antigen (PSA) level exceeding 4 ng/mL, a prostate volume exceeding 40 ml, an amount of remaining urine of 300 mL or more, the utilize of 5-alpha reductase inhibitors (5-ARIs) in the past three months, a history of prostate surgery or malignancy, urethral stricture, urinary retention, bladder stones, neurological diseases affecting bladder function, cardiovascular diseases, and treatment with nitrates.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
IPSS (International Prostate Symptom Score) | at presentation, 1,3 and 6 month after treatment
  The International Prostate Symptom Score (IPSS) is a questionnaire used to assess the severity of symptoms related to the lower urinary tract, often associated with conditions like benign prostatic hyperplasia (BPH) in men. It helps healthcare providers determine the severity of symptoms, monitor changes over time, and guide treatment decisions.
  The IPSS consists of 8 questions, covering symptoms such as:
  Incomplete Emptying: Feeling that the bladder is not fully emptied after urination.
  Frequency: How often you feel the need to urinate. Intermittency: Whether urine flow starts and stops during urination. Urgency: How urgently you need to urinate. Weak Stream: The strength of the urine stream. Straining: How much effort is needed to urinate. Nocturia: How many times you wake up at night to urinate. Quality of Life: General assessment of how urinary symptoms affect your quality of life.
  Each question is rated on a scale from 0 (no symptoms) to 5

SECONDARY OUTCOMES:
IIEF-5 (five-item International Index of Erectile Function) | at presentation, 1,3 and 6 month after treatment
  The Five-Item International Index of Erectile Function (IIEF-5) is a short, standardized questionnaire used to assess erectile function in men. It is often used to screen for erectile dysfunction (ED) and can help determine its severity.
  The IIEF-5 consists of 5 questions related to the ability to achieve and maintain an erection, as well as overall satisfaction with sexual activity. The questions are scored on a scale from 0 to 5, with a higher score indicating better erectile function.
  Here are the five questions:
  How often have you had erections during sexual activity? Scale: 0 (Almost never or never) to 5 (Almost always or always) When you had erections with sexual stimulation, how often were your erections hard enough for penetration? Scale: 0 (Almost never or never) to 5 (Almost always or always) During sexual activity, how often were you able to maintain your erection after you had penetrated? Scale: 0 (Almost never or never) to 5 (Almost always or always) How satisfied have
Q-max (maximum urinary flow rate) | at presentation, 1,3 and 6 month after treatment
  The maximum urinary flow rate (Qmax) refers to the highest rate at which urine is expelled from the bladder during urination. It is commonly measured during a uroflowmetry test, which is a diagnostic procedure used to evaluate the efficiency of the urinary system.
  How it's measured:
  A person is asked to urinate into a device that records the volume and flow rate of urine over time.
  The test measures the peak flow rate, which is the fastest rate at which urine is being passed during the process.
  It's typically expressed in milliliters per second (mL/s).
  What the results mean:
  Normal Qmax: For men, a typical normal maximum urinary flow rate is usually between 15 and 25 mL/s. In women, normal values can range slightly, depending on factors like age, but are often similar.
  Low Qmax: A flow rate lower than normal could indicate an obstruction or narrowing in the urinary tract, bladder dysfunction, or conditions such as benign prostatic hyperplasia (BPH) in men or pelvic floor dysfunctio
PVR (post-void residual urine) | at presentation, 1,3 and 6 month after treatment
  it is a measure of post-void residual urine in bladder using ultrasound
QoL (quality of life) | at presentation, 1,3 and 6 month after treatment
  The QoL Question:
  In the IPSS, there is a single question that asks:
  "If you were to spend the rest of your life with your urinary condition, how would you feel about that?"
  Patients rate their quality of life on a scale from 0 to 6, where:
  0 = "Delighted"
  1. = "Pleased"
  2. = "Mostly satisfied"
  3. = "Mixed"
  4. = "Mostly dissatisfied"
  5. = "Very dissatisfied"
  6. = "Terrible" This score helps healthcare providers understand how bothersome the symptoms are, and it contributes to determining the need for treatment.
  Significance of the QoL Score:
  Low QoL Score (0-2): Indicates that the patient is generally satisfied with their condition or feels only mild disruption to their life. This might suggest that treatment isn't urgently needed, or that the symptoms are not significantly affecting their daily activities.
  Moderate QoL Score (3-4): Suggests that the symptoms are having a moderate impact on daily life, and treatment may be considered to alleviate the burden.
  High QoL Score (5-6): Indica

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Mahmoud Dogha, Al Fayyum, Fayoum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] MacDonald R, Brasure M, Dahm P, Olson CM, Nelson VA, Fink HA, Risk MC, Rwabasonga B, Wilt TJ. Efficacy of newer medications for lower urinary tract symptoms attributed to benign prostatic hyperplasia: a systematic review. Aging Male. 2019 Mar;22(1):1-11. doi: 10.1080/13685538.2018.1434503. Epub 2018 Feb 2. PMID 29394114
- [Background] Morton A, Williams M, Perera M, Teloken PE, Donato P, Ranasinghe S, Chung E, Bolton D, Yaxley J, Roberts MJ. Management of benign prostatic hyperplasia in the 21st century: temporal trends in Australian population-based data. BJU Int. 2020 Sep;126 Suppl 1:18-26. doi: 10.1111/bju.15098. Epub 2020 Jun 17. PMID 32558340
- [Background] Yamanishi T, Kaga K, Sakata K, Yokoyama T, Kageyama S, Fuse M, Tokunaga S. A randomized controlled study of the efficacy of tadalafil monotherapy versus combination of tadalafil and mirabegron for the treatment of persistent overactive bladder symptoms in men presenting with lower urinary tract symptoms (CONTACT Study). Neurourol Urodyn. 2020 Feb;39(2):804-812. doi: 10.1002/nau.24285. Epub 2020 Jan 21. PMID 31961963
- [Background] Michel MC, Vrydag W. Alpha1-, alpha2- and beta-adrenoceptors in the urinary bladder, urethra and prostate. Br J Pharmacol. 2006 Feb;147 Suppl 2(Suppl 2):S88-119. doi: 10.1038/sj.bjp.0706619. PMID 16465187
- See also: EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. — https://pubmed.ncbi.nlm.nih.gov/25613154/
- See also: Efficacy of newer medications for lower urinary tract symptoms attributed to benign prostatic hyperplasia: a systematic review. Aging Male. — https://pubmed.ncbi.nlm.nih.gov/29394114/
- See also: Management of benign prostatic hyperplasia in the 21st century: temporal trends in Australian population-based data. — https://pubmed.ncbi.nlm.nih.gov/32558340/
- See also: A randomized controlled study of the efficacy of tadalafil monotherapy versus combination of tadalafil and mirabegron for the treatment of persistent overactive bladder symptoms in — https://pubmed.ncbi.nlm.nih.gov/31961963/
- See also: Alpha1-, alpha2- and beta-adrenoceptors in the urinary bladder, urethra and prostate. — https://pubmed.ncbi.nlm.nih.gov/16465187/